**Project Title:** Improving Community Ambulation for Stroke Survivors using Powered Hip Exoskeletons with Adaptive Environmental Controllers

NCT Number: NCT03924752

Date: November 17, 2021

## **Statistical Analysis Plan**

Means of the subject's self-selected walking speed for all different locomotion modes (level-ground, ramp ascent, ramp descent, stair ascent, and stair descent) for all assistance conditions (no exoskeleton and exoskeleton with assistance) across 10 subjects were computed. We performed a two-way repeated measures analysis of variance (locomotion mode and assistance type as independent variables) on the subject's walking speed by setting an  $\alpha$  value to 0.05 (MATLAB 2021b, Mathworks, USA).